CLINICAL TRIAL: NCT06775795
Title: The Bioavailability of Iodine in Plant-based Milk Alternatives
Acronym: IoBIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FHMS 23-24 161 EGA
Record Dates: First submitted 2025-01-03; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Iodine Deficiency
Keywords: iodine bioavailability; iodine; milk; plant-based
MeSH Terms: interventions — Soy Milk; Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cow's milk (Active Comparator): Semi-Skimmed UHT Milk (estimated iodine concentration: 350 µg/L) providing approximately 200 µg of iodine (approx. 570mL).
  Interventions: Dietary Supplement: Cow's milk
- Oat milk alternative (Experimental): Oat Drink (estimated iodine concentration: 370 µg/L) providing approximately 200 µg of iodine (approx. 545mL).
  Interventions: Dietary Supplement: Oat milk
- Soya milk alternative (Experimental): Soya Drink (estimated iodine concentration: 460 µg/L) providing approximately 200 µg of iodine (approx. 435mL).
  Interventions: Dietary Supplement: Soya milk

INTERVENTIONS:
Dietary Supplement: Oat milk — Participants will consume one portion of plant-based milk alternative (oat) which will provide approximately 200 µg of iodine
  Arms: Oat milk alternative
Dietary Supplement: Soya milk — Participants will consume one portion of plant-based milk alternative (soya) which will provide approximately 200 µg of iodine
  Arms: Soya milk alternative
Dietary Supplement: Cow's milk — Participants will consume one portion of semi-skimmed cow's milk which will provide approximately 200 µg of iodine
  Arms: Cow's milk

SUMMARY:
Iodine is a mineral commonly found in seafood and dairy products such as milk and cheese. Iodine is important as it is required to make thyroid hormones which regulate growth and metabolism at all stages of life. The UK population has been iodine-sufficient for many years, however, there is now concern that iodine deficiency may be more prevalent than previously thought. This is a concern because iodine deficiency during pregnancy can result in cognitive impairment and developmental delays in children.

This study will to measure the ability to absorb iodine from plant-based milk alternatives fortified with iodine and compare with cow's milk in adults. Knowing the actual iodine bioavailability from plant-based alternatives is important because plant-based milk alternatives are becoming increasingly popular, especially in young adults, and are used as a replacement for cow's milk.

In this study, participants will consume three test drinks (cow's milk, soya milk and oat milk), one per week. The study will start with the cows' milk and the other two drinks will be administered in a random order with a crossover design. We will ask participants to follow a low iodine diet for three days leading up to the test day where they will drink one of the test drinks. Participants will then keep a food diary and collect their urine for the following 24 hours. Participants will then go back to their usual diet for at least four days before starting the next arm of the study with another test drink. This data will be used to calculate how much iodine was absorbed.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported healthy adults
* Aged 18+
* English speakers
* Signed consent form
* No allergies or intolerances to the study drinks
* Not following a vegan diet (participants will be required to drink cow's milk)

Exclusion Criteria:

* Pregnancy or lactating (according to the participants own statement)
* Living outside of the UK
* Involvement in another research study where diet is restricted or modified
* History of thyroid disease (according to the participants own statement)
* Any metabolic, gastrointestinal or chronic disease such as diabetes, hepatitis, hypertension, or cancer (according to the participants own statement)
* Use of iodine containing supplements within 1 week prior to study start
* Inadequate (<70 µg/day) or excessive (>500 µg/day) iodine intake from food (assessed during screening with previously validated iodine-specific FFQ)
* Use of iodine-containing disinfectants (betadine)
* Exposure to iodine-containing X-ray/ computed tomography contrast agent within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Urinary iodine excretion | A single spot-urine sample collected on days: 2, 9, 16 Urine collected for 24 hours after consumption of test drink on days: 3, 10, 17
  1 sport urine sample will be collected the day before test drink consumption and a 24-hour urine sample will be collected following the test drink consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No